CLINICAL TRIAL: NCT03250065
Title: Development of the "Sensing Endotracheal Tube": an Optical Multi-parameter Monitoring System.
Brief Title: The Sensing ET Tube
Acronym: SETT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: City, University of London (Other)
Collaborators: Barts & The London NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RCBE/2015/01
Record Dates: First submitted 2017-08-09; First posted 2017-08-15 (Actual); Last update posted 2018-02-12 (Actual); Status verified 2018-02

CONDITIONS: Diagnostic Equipment; Oximetry; Pulse Rate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ETT Study Group (Experimental): The Sensing ET Tube study Group
  Interventions: Device: Application of prototype sensor to a standard endotracheal tube

INTERVENTIONS:
Device: Application of prototype sensor to a standard endotracheal tube — During anaesthesia the device under study, a prototype saturation sensor will be applied to a standard endotracheal tube that ventilates the patient as normal.

SUMMARY:
This proposal describes the development of a 'Sensing ET Tube'. This device will replace the standard endotracheal (ET) tube used in anaesthesia and in ventilated intensive care patients and provide key vital signs monitoring utilising optoelectronic sensors. Continuous monitoring of patients' arterial oxygen saturation is essential during surgery, however pulse oximeters often misread or fail altogether as a result of peripheral vasoconstriction, hypotension or hypovolaemia. The Sensing ET Tube will allow continuous measurement of oxygen saturation and other parameters, such as pulse rate, from a single internal site, and will reduce the number of surface sensors placed on the skin and the number of electrical connections to the patient. The applicants have already developed similar sensor technology in the oesophagus and other internal locations. A pilot clinical evaluation of the device will be completed in anaesthetised patients undergoing surgery. The project will lead to further development of a multi-sensor tracheal platform for comprehensive anaesthesia and intensive care monitoring.

DETAILED DESCRIPTION:
The aim of this project is to develop and evaluate a novel medical device known as the 'Sensing ET Tube' for measuring oxygen levels in patients undergoing surgical operations. The device replaces the standard breathing tube used in surgery and incorporates photonic sensors for measurement of the patient's oxygen level and other vital signs. Currently this information is supplied from finger probes, which can fail often, for example when the patient is cold or when the blood pressure is low. The new device is completely harmless and allows the anaesthetist to monitor the oxygen level from the central region of the body using minimal connections. If successful, future work is planned to incorporate other sensors into the system, providing a complete overview of the health of the patient. This will greatly simplify the process of patient monitoring while reducing the number of failures, improving patient safety and reducing operating costs.

A clinical trial is planned in up to 50 patients undergoing general anaesthesia, which will quantitatively evaluate the accuracy and reliability of the measured clinical variables and the device's expected performance in mainstream operation. This information will provide the basis for further commercial development, most likely through partnership with a medical device manufacturer.

To summarise, the main aims of the project are:

* Investigate photoplethysmographic signals from the human trachea and identify viability to measure heart rate, and blood oxygen saturation by comparison with "gold standard" techniques.
* Evaluate custom-designed endotracheal sensor for operation and determine ideal electrical characteristics for optimal operation (current supply, detector amplification etc.)

ELIGIBILITY:
Inclusion Criteria:

* ASA I-III
* 18 Years and older
* Undergoing elective surgery requiring general anaesthesia, and endotracheal tube as part of their anaesthetic.

Exclusion Criteria:

* Those who refuse consent
* Known or potentially difficult airway
* Respiratory conditions including severe asthma, COPD, lung cancer etc.
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2017-03-03 (Actual); Primary Completion 2017-07-31 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
To validate the pulse oximetry signals from the trachea during anaesthesia for their suitability in determining vital signs, not limited to just oxygen saturation. | 1 year
  Raw optical electrical signals related to the absorbion of red and infrared light from the prototype sensor by the tissue in the trachea will be assessed for their viability to reliable determine pulse rate and oxygen saturation compared to the standard clinical devices during surgery. The signals will be further analysed to look for correlation with recorded blood pressure measurents and respiration rates.

CONTACTS AND LOCATIONS:
Overall Officials: Saowarat Snidvongs, MD, Principal Investigator — Barts and The London NHS Trust; Justin Phillips, PhD, Study Director — City, University of London; Panayiotis A Kyriacou, PhD, Study Chair — City, University of London
Locations (2):
- United Kingdom (2):
  - City, University of London, London
  - Barts and The London NHS Trust, London

IPD SHARING:
Plan to Share IPD: No
all data is anonymised and raw signals are only shared among the named investigators